CLINICAL TRIAL: NCT04265326
Title: Validity and Reliability of the Turkish Version of the Head and Neck Cancer Inventory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Head of Geriatric Rehabilitation Department, Izmir Bakircay University
Other Study IDs: 2018-146
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer patients: Turkish patients diagnosed with Head and Neck Cancer
  Interventions: Other: Measurement of Quality of Life

INTERVENTIONS:
Other: Measurement of Quality of Life — Quality of life will be measured using Head and Neck Cancer Inventory and The Functional Assessment of Cancer Therapy - Head and Neck Cancer Version 4

SUMMARY:
The primary treatment option of many patients with head and neck cancer is surgery, radiotherapy and chemotherapy. In the literature, functional problems that occur after surgical interventions applied to head and neck cancer patients are frequently mentioned. Morbidities resulting from the combined application of radiotherapy and chemotherapy are based on more anecdotal information and critical data on long-term functional outcomes in this patient group are scarce. The aim of this study is to make the validity, reliability and cultural adaptation of the Head and Neck Cancer Inventory in Turkish.

DETAILED DESCRIPTION:
In the literature, there are general cancer scales developed to evaluate the quality of life of head and neck cancer patients and sub scales associated with head and neck cancers developed in addition to these scales. In addition, scales specific to head and neck cancers have also been developed. However, previous research shows that even general health status scales or cancer-specific scales cannot determine outcomes related to many head and neck cancer patients. In addition, items containing multiple functions and patients' attitudes (behaviors) cannot be analyzed separately in any of the scales specific to head and neck cancer. Very few surveys contain items related to patients' attitudes (behaviors), or the number of items related to this topic is small because most of these scales are functional items. Unlike its counterparts in the literature, Head and Neck Cancer Inventory evaluates the attitudes (behaviors) of patients associated with various functions in daily life. Head and Neck Cancer Inventory is the only scale in the literature that contains the basic features of the health conditions declared by the patient and has been developed specifically for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting to participate in the study
* Patients whose native language is Turkish
* Patients diagnosed with head and neck cancer

Exclusion Criteria:

* Patients whose health conditions are too bad to fill the scale
* Having a serious mental disorder or dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Turkish patients diagnosed with head and neck patients
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Head and Neck Cancer Inventory | At baseline
  It is a scale consisting of 30 items in total, containing 4 main categories [speech (10 items), eating (10 items), aesthetics (2 items), social disorders (7 items)] evaluating the quality of life related to head and neck cancer and an additional item evaluating the overall quality of life. This inventory reflects both functionality (how functional the patient is) and attitudes (how satisfied is the patient's functional level) using a 5-point Likert-type scale. This scale does not have a summary score representing all items, the score of 4 different categories can be calculated. The higher the scores, the better the quality of life [2].

SECONDARY OUTCOMES:
The Functional Assessment of Cancer Therapy - Head and Neck Cancer Version 4 | At baseline
  In addition to the 27-item Cancer Treatment Functional Evaluation-General (FACT-G) scale, this scale consists of 9 additional items specific to head and neck cancer. FACT G consists of 4 main categories that evaluate physical (7 items), social (7 items), emotional (6 items) and functional status (7 items). Each item is scored by patients with a Likert type classification ranging from 0 (none) to 4 (too many). Points are calculated separately for each category. A summary score is also calculated for FACT-G and total FACT-H & N [3]. The questionnaire is available in Turkish version [9].

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Cohen EE, LaMonte SJ, Erb NL, Beckman KL, Sadeghi N, Hutcheson KA, Stubblefield MD, Abbott DM, Fisher PS, Stein KD, Lyman GH, Pratt-Chapman ML. American Cancer Society Head and Neck Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 May;66(3):203-39. doi: 10.3322/caac.21343. Epub 2016 Mar 22. PMID 27002678
- [Background] Funk GF, Karnell LH, Christensen AJ, Moran PJ, Ricks J. Comprehensive head and neck oncology health status assessment. Head Neck. 2003 Jul;25(7):561-75. doi: 10.1002/hed.10245. PMID 12808660
- [Background] Heutte N, Plisson L, Lange M, Prevost V, Babin E. Quality of life tools in head and neck oncology. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Feb;131(1):33-47. doi: 10.1016/j.anorl.2013.05.002. Epub 2013 Nov 28. PMID 24291153
- [Background] Gliklich RE, Goldsmith TA, Funk GF. Are head and neck specific quality of life measures necessary? Head Neck. 1997 Sep;19(6):474-80. doi: 10.1002/(sici)1097-0347(199709)19:63.0.co;2-w. PMID 9278754
- [Background] D'Antonio LL, Zimmerman GJ, Cella DF, Long SA. Quality of life and functional status measures in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 1996 May;122(5):482-7. doi: 10.1001/archotol.1996.01890170018005. PMID 8615964
- [Background] List MA, D'Antonio LL, Cella DF, Siston A, Mumby P, Haraf D, Vokes E. The Performance Status Scale for Head and Neck Cancer Patients and the Functional Assessment of Cancer Therapy-Head and Neck Scale. A study of utility and validity. Cancer. 1996 Jun 1;77(11):2294-301. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-S. PMID 8635098
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568